CLINICAL TRIAL: NCT07092722
Title: A Randomized, Double Blind, Placebo Controlled Parallel Arm Clinical Study to Evaluate the Efficacy of LN18178 in Improving Muscle Strength, Aerobic Capacity and Body Composition in Healthy Young Males
Brief Title: Efficacy of LN18178 in Improving Muscle Strength, Aerobic Capacity and Body Composition in Healthy Young Males
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GENCOR Lifestage Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GNC/MS/LN18178/25; CTRI/2025/07/091371 (Registry Identifier: Clinical Trial Registry - India Board)
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Muscle Strength Recovery; Endurance; Healthy Human Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LN18178 (Experimental): 400 mg, One capsule to be consumed in the morning after breakfast with water for 12 Weeks
  Interventions: Dietary Supplement: LN18178
- Placebo (Other): One capsule to be consumed in the morning after breakfast with water for 12 Weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LN18178 — 400 mg, One capsule to be consumed in the morning after breakfast with water for 12 Weeks
  Arms: LN18178
Dietary Supplement: Placebo — One capsule to be consumed in the morning after breakfast with water for 12 Weeks
  Arms: Placebo

SUMMARY:
The Purpose of the study is to evaluate the efficacy of LN18178 in improving muscle strength, aerobic capacity and body composition in healthy young males.

DETAILED DESCRIPTION:
A total of 120 male subjects aged between 36 and 50 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either LN18178:400 mg or Placebo at 1:1 ratio. The subjects will be instructed to take one capsule daily in the morning after breakfast with water for 12 weeks. Apart from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition safety and tolerability. The safety assessment of the LN18178 will also include routine laboratory investigations on blood, urine and clinical chemistry at screening and the final visit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Untrained healthy male subjects aged between 36 and 50 years with a Body Mass Index (BMI) between 22 and 27 kg/m2.
2. Willingness to do exercise training program during the course of the study.
3. Subject considered generally healthy as per health history and routine clinical investigations.
4. Ability to understand the risks and benefits of the protocol.
5. Subject should provide written informed consent and agree to be available for regular follow up throughout the study duration.
6. Subjects who are sexually active must agree to use adequate non-hormonal contraception during the study
7. Subjects agree to maintain current diet and activity level.
8. Subject agrees not to start any new therapies for energy boosting supplements or protein supplements or health drinks during the course of the study.
9. Subjects willing to refrain from drinking coffee or caffeinated drinks or beverages during the study.

Exclusion Criteria:

1. Subjects who are resistance trained or undergoing resistance training.
2. Subjects with blood pressure more than or equal to 140/90 mmHg, fasting plasma glucose more than 125 mg/dL and abnormal ECG.
3. Subjects underwent treatment for COVID-19 within last 3 months or tested positive during the study will be excluded.
4. Evidence or history of musculoskeletal, respiratory, haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic diseases, malignancies.
5. Subjects diagnosed with sleep apnea or related disorders.
6. Subjects consuming medications that can interfere with muscle mass such as corticosteroids, testosterone replacement or anabolic drugs.
7. History of psychiatric disorder that may impair the ability of subjects to provide written informed consent.
8. Subjects consuming alcohol (more than 3 standard drinks per week) or smokers ( more than 3 cigarettes per day).
9. Subjects who consume recreational drugs (such as cocaine, methamphetamine, marijuana, etc.) or chewable tobacco products.
10. Subjects under medications including anti-hypertensives, antidepressants, anticholinergics, inhaled beta agonists, anti-hyperlipidemics, psychotropics etc.
11. Subjects using any centrally acting anorectic agents, drugs that inhibit the absorption of nutrients and endocannabinoid neuromodulators during the two weeks prior to enrolment into the study.
12. Subjects who underwent major surgical procedures in last 6 months.
13. Subject with HIV positive or history of any other STDs.
14. Subject has participated in a clinical study within the last 30 days prior to recruitment or concurrently participating in another study

    -

Ages: 36 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Untrained healthy male subjects
Enrollment: 120 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle strength (1-RM leg press) | Week 0, Week 2, Week 4, Week 8 and Week 12
  It's the maximum amount of weight a subject can lift for one repetition of leg press. As the weight lifted increases, muscle strength also rises

SECONDARY OUTCOMES:
Change in Muscle strength ( 1-RM bench press) | Week 0, Week 2, Week 4, Week 8 and Week 12
  It's the maximum amount of weight a subject can lift for one repetition of bench press. As the weight lifted increases, so does muscle strength.
Change in Muscle endurance (Repetitions to failure for leg press and bench press using 80% 1RM) | Week 0, Week 2, Week 4, Week 8 and Week 12
  It refers to the maximum number of repetitions a person can perform at 80% of their one-repetition maximum (1RM) weight on the leg press and bench press. An increase in repetitions reflects improved muscle endurance.
Change in training volume/capacity | Week 0, Week 2, Week 4, Week 8 and Week 12
  It is a calculated value obtained by multiplying the number of sets, the number of repetitions per set, and the weight lifted in kilograms for an exercise. As training volume increases, so does muscle strength.
Change in VO2 max testing (graded exercise test while O2 consumption measured) | Week 0 and Week 12
  The maximum amount of oxygen the body utilizes during graded exercise on an ergometer is measured as VO₂ max. An increase in VO2 max indicates improved cardiovascular fitness
Change in Lean body mass (DEXA) | Week 0 and Week 12
  A low-dose X-ray (DEXA) is used to measure a person's lean mass. An increase in lean mass signifies notable improvements in muscle development.
Change in Rate of Perceived Exertion (RPE) using 6-20 point Borg scale for exercise intensity | Week 0, Week 2, Week 4, Week 8 and Week 12
  It is a measure of how much exertion a person feels at the end of an exercise session. A decrease in ratings on the Borg scale indicates reduced perceived exertion, reflecting improvements in muscle strength and endurance.
Change in subjective rating of Energy, Fatigue, Focus and Confidence using VAS | Week 0, Week 2, Week 4, Week 8 and Week 12
  The Visual Analogue Scale (VAS) is a 100 mm line, with zero representing the minimum score and 100 representing the maximum. Higher ratings on the scale correspond to increased levels of energy, reduced fatigue, and greater focus and confidence
Change in subjective feeling of mental acuity, concentration, calmness and quality of sleep using VAS | Week 0, Week 2, Week 4, Week 8 and Week 12
  The Visual Analogue Scale (VAS) is a 100 mm line, where zero represents the minimum score and 100 the maximum. Higher ratings on the scale indicate greater mental acuity, improved concentration, increased calmness, and better quality of sleep."
Change in Physical Activity Enjoyment Scale-8 (PACES) | Week 0, Week 2, Week 4, Week 8 and Week 12
  The Physical Activity Enjoyment Scale-8 uses a 7-point bipolar rating scale to assess how a person currently feels about the physical activity they have been performing. Higher total scores indicate greater enjoyment of the activity.
Change in Serum biomarkers (IGF-1 - Insulin-like growth factor-1) | Week 0 and Week 12
  Insulin-like Growth Factor 1 (IGF-1) is a hormone that plays a key role in promoting muscle growth in adults. As serum IGF-1 levels increase, there is a corresponding rise in lean muscle mass
Change in Serum biomarkers Myostatin | Week 0 and Week 12
  Myostatin is a myokine produced by muscle cells that serves as a negative regulator of muscle growth. Higher serum myostatin levels are associated with reduced lean mass and decreased muscle strength.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandit SL, Yaligar D, Halemane M, Bhat A. A proprietary blend of standardized Punica granatum fruit rind and Theobroma cocoa seed extracts mitigates aging males' symptoms: A randomized, double-blind, placebo-controlled study. Int J Med Sci. 2022 Jul 11;19(8):1290-1299. doi: 10.7150/ijms.73645. eCollection 2022. PMID 35928723
- [Background] Sreeramaneni PGA, Yalamanchi A, Konda MR, Cherukuri SHV, Maroon JC. A Proprietary Herbal Blend Containing Extracts of Punica granatum Fruit Rind and Theobroma cocoa Seeds Increases Serum Testosterone Level in Healthy Young Males: A Randomized, Double-Blind Placebo-Controlled Study. J Diet Suppl. 2023;20(3):411-427. doi: 10.1080/19390211.2022.2035037. Epub 2022 Feb 6. PMID 35129040
- [Background] Rawson ES, Volek JS. Effects of creatine supplementation and resistance training on muscle strength and weightlifting performance. J Strength Cond Res. 2003 Nov;17(4):822-31. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 14636102
- [Background] Garcia-Hermoso A, Sanchez-Lopez M, Martinez-Vizcaino V. Effects of Aerobic Plus Resistance Exercise on Body Composition Related Variables in Pediatric Obesity: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pediatr Exerc Sci. 2015 Nov;27(4):431-40. doi: 10.1123/pes.2014-0132. Epub 2015 Apr 22. PMID 25902557
- [Background] Ramos-Campo DJ, Andreu Caravaca L, Martinez-Rodriguez A, Rubio-Arias JA. Effects of Resistance Circuit-Based Training on Body Composition, Strength and Cardiorespiratory Fitness: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Apr 28;10(5):377. doi: 10.3390/biology10050377. PMID 33924785
- [Background] Holloszy JO. The biology of aging. Mayo Clin Proc. 2000 Jan;75 Suppl:S3-8; discussion S8-9. PMID 10959208
- [Background] Suchomel TJ, Nimphius S, Stone MH. The Importance of Muscular Strength in Athletic Performance. Sports Med. 2016 Oct;46(10):1419-49. doi: 10.1007/s40279-016-0486-0. PMID 26838985
- [Background] Kell RT, Bell G, Quinney A. Musculoskeletal fitness, health outcomes and quality of life. Sports Med. 2001;31(12):863-73. doi: 10.2165/00007256-200131120-00003. PMID 11665913